CLINICAL TRIAL: NCT01180218
Title: Comparison of Complete Lesion Versus Culprit Lesion Revascularization in Acute ST Elevation Myocardial Infarction Patients With Multivessel Disease Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Complete Lesion Versus Culprit Lesion Revascularization
Acronym: COCUA
Status: Temporarily not available | Type: Expanded Access
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seung Woon Rha, Associate professor, Korea University Guro Hospital
Other Study IDs: KoreaUGuroH_1
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Myocardial Infarction
Keywords: myocardial revascularization; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Procedure: complete revascularization — -Complete revascularization : one time primary percutaneous coronary intervention (PCI) of the culprit and nonculprit lesions in patient with ST elevateion myocardial infarction (STEMI) and multivessle disease
Procedure: Culprit revasularization — Culprit revascularization : PCI of only the culprit lesion and staged nonculprit PCI at a later date in patients with ST-segment elevation myocardial infarction (STEMI) and multivessel disease.

SUMMARY:
To investigate the clinical outcomes of acute myocardial infarction (AMI) patients with multivessel disease undergoing percutaneous coronary intervention (PCI) either in infarct-related artery only or in multivessel in Drug eluting stents (DES) era, using the everolimus-eluting stent (Promus™ Element™ Stent, Boston Scientific) in real-world clinical practice.

DETAILED DESCRIPTION:
Acute ST segment elevation myocardial infarctions (STEMI) is a systemic prothrombotic milieu, often involves more than one coronary artery, even though it predominantly affects plaque rupture and its consequences in one coronary artery territory (culprit artery territory)(1). Also, Multivessel disease (MVD), a well known predictor of poor clinical outcomes occurs in acute myocardial infarction (AMI) patients (pts) between 40% and 65%(2, 3).

In acute STEMI, achieving the maximum myocardial reperfusion and salvage by primary percutaneous intervention of culprit lesion is the preferred reperfusion strategy as per the latest ACC/AHA and ESC guidelines(4, 5). At presently there is no consensus regarding the management of significant non culprit lesions during the initial presentation in hemodynamically stable STEMI pts(6, 7).Although multivessel revascularization seems to improve the myocardial reperfusion and its salvage by limiting infarct size, improving ejection fraction (EF) and stabilizing the vulnerable plaques in acute AMI presentation, revascularization of non IRAs yielded conflicting results in the BMS era(2, 7-13). Balancing the above merits with increased risk of having higher periprocedural MI due to multivessel stent implantations in non IRAs are paramount importance in deciding the revascularization strategy in MVD STEMI pts(13-15). Drug eluting stents (DES) implantations after primary PCI are increasing in the real world scenario after the establishment of its safety by the multiple Meta analyses and few randomized trials(16-19).Even though DES reduces recurrent revascularizations in acute STEMI pts, the merits and demerits of its usage in treating non IRAs in multivessel disease pts with STEMI are largely unknown in this modern PCI era(16, 19). The aim of the study was to compare the clinical outcomes between culprit lesion revascularization (CLR) group and complete revascularization (CR) group where CR group includes treatment of both IRA and non IRAs) strategy in MVD STEMI pts in the real world scenario utilizing DES.

Primary percutaneous coronary intervention (PCI) is established as the treatment of choice for acute ST segment elevation myocardial infarction (STEMI). During the procedure, the culprit artery recanalization allows reperfusion of the myocardium and improves healing of the injured tissue (20, 21). Recent studies showed that in the AMI setting, the pathophysiology involves the whole coronary artery tree (21), and nearly 40% to 65% patients presenting with AMI have multivessel disease (22), (23), (24), (25) and plaque instability might develop in a multifocal pattern, resulting in unstable plaques in anatomically remote locations and may emerge as the cause of recurrent acute coronary syndrome. Current guidelines of primary PCI recommend treating the culprit vessel in the urgent procedure, leaving the other untreated vessels to another elective procedure. Multivessel PCI is recommended only for patients with cardiogenic shock (20, 21, 26). By this strategy, the operator intends to avoid the potential procedural complications that may deteriorate the patient's left ventricular function and clinical condition during acute myocardial infarction. Therefore, only few reports describe the results of simultaneous non culprit vessel PCI for patients undergoing mechanical reperfusion for STEMI.

An early study of primary PCI for patients with multivessel disease showed favorable results with a strategy of staged percutaneous revascularization after acute recanalization of the culprit artery (24). In recent years with the use of stents and platelet glycoprotein IIb/IIIa inhibitors, the outcome of elective multivessel PCI has markedly improved (27, 28). More recent reports on simultaneous percutaneous revascularization of non-culprit arteries indicate that this may be a good strategy for patients with AMI found to have multivessel disease during primary angioplasty (29). According to some studies involving Coronary artery bypass graft (CABG) surgery, complete revascularization showed to be associated with better outcomes as compared with incomplete revascularizations (30), (31). In the Bare Metal Stent (BMS) era, long term event free survival rates of patients undergoing primary intervention for multivessel disease was shown to be as low as 48.5% (32). In-Stent Restenosis was seen as one of the major drawback which varied from 8% to as high as 80% at 6 months, according to both anatomic and clinical risk factors (33). However, introduction of Drug Eluting Stent (DES) showed promising results and similar results with either PCI with DES or CABG for patients with multivessel disease were seen(34), (35), [12].

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject is able to verbally confirm understandings of risks, benefits and treatment of culprit or complete revascularization using everolimus eluting coronary stent (Promus™ Element™ Stent) and he or she or his or her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject must have significant more than two target lesions and requiring primary PCI for acute ST elevation myocardial infarction (STEMI) within 48hrs
* Target lesion(s) must be located in a native coronary artery with visually estimated diameter of less than 2.5 mm and more than 4.0 mm.
* Target lesion(s) must be amenable for percutaneous coronary intervention

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications:

Heparin Aspirin Both Clopidogrel and Ticlopidine Everolimus Platinum chromium Contrast media

* Patients with documented sensitivity to contrast media which can be effectively pre medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.
* Systemic (intravenous) everolimus use within 12 months. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* History of bleeding diathesis or known coagulopathy (including heparin- Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months,induced thrombocytopenia), or will refuse blood transfusions.
* An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first 6 months post enrollment.
* Non-cardiac comorbid conditions are present with life expectancy over 1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* Patients with more than 25 percentage of LVEF or those with cardiogenic shock
* Creatinine level more than 3mg per dL or dependence on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Seung Woon Rha, Principal Investigator — professor
Locations (1):
- Seung Woon Rha, Seoul, South Korea

REFERENCES:
- [Result] Vlaar PJ, Mahmoud KD, Holmes DR Jr, van Valkenhoef G, Hillege HL, van der Horst IC, Zijlstra F, de Smet BJ. Culprit vessel only versus multivessel and staged percutaneous coronary intervention for multivessel disease in patients presenting with ST-segment elevation myocardial infarction: a pairwise and network meta-analysis. J Am Coll Cardiol. 2011 Aug 9;58(7):692-703. doi: 10.1016/j.jacc.2011.03.046. PMID 21816304
- [Derived] Park S, Rha SW, Choi BG, Cho JH, Park SH, Lee JB, Kim YH, Park SM, Choi JW, Park JY, Shin ES, Lee JB, Suh J, Chae JK, Choi YJ, Jeong MH, Cha KS, Lee SW, Kim U, Kim GC, Choi WG, Cho YH, Cho DK, Ahn J, Suh SY, Choi SY, Byun JK, Cha JA, Hyun SJ, Kim JB, Choi CU, Park CG. Immediate versus staged complete revascularization in patients with ST-segment elevation myocardial infarction and multivessel coronary artery disease: results from a prematurely discontinued randomized multicenter trial. Am Heart J. 2023 May;259:58-67. doi: 10.1016/j.ahj.2023.01.020. Epub 2023 Feb 7. PMID 36754106